CLINICAL TRIAL: NCT01606748
Title: An Open-Label, Non-controlled, Non-randomized Sequential Design, Drug-Interaction Study of Necitumumab (IMC-11F8) in Combination With Gemcitabine-Cisplatin in Patients With Advanced Solid Cancers
Brief Title: A Drug-Interaction Study of Necitumumab (IMC-11F8) in Combination With Gemcitabine-Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14473; CP11-1115 (Other: ImClone Systems); I4X-IE-JFCJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Malignant Solid Tumor
Keywords: Advanced Malignant Solid Tumors; Solid Cancers; Non-small Cell Lung Cancer; NSCLC; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — necitumumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Necitumumab, Gemcitabine and Cisplatin (Experimental): The study will be conducted in two sequential periods: a 3-week PK run-in participants will be treated sequentially with single doses of cisplatin, gemcitabine, and necitumumab. Cycle 1 will begin immediately following the PK run-in period.
  Interventions: Biological: Necitumumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Necitumumab — PK Run-In Period: Necitumumab administered on Day 3 of the 3-week PK run-in period as an intravenous (I.V.) infusion at an absolute dose of 800 mg
  Treatment Cycles: Necitumumab administered on Days 1 and 8 of every 3-week cycle as an intravenous (I.V.) infusion at an absolute dose of 800 mg
  Participants in Cohort 1 will receive necitumumab Process C drug product and participants in Cohort 2 will receive necitumumab Process D drug product
  Other Names: IMC-11F8; LY3012211
Drug: Gemcitabine — PK Run-In Period: Gemcitabine administered on Day 1 of the 3-week PK run-in period as an I.V. infusion at a dose of 1250 milligram per square meter (mg/m2)
  Treatment Cycles: Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an I.V. infusion at a dose of 1250 mg/m2
  Other Names: Gemzar®; LY188011
Drug: Cisplatin — PK Run-In Period: Cisplatin administered on Day 1 of the 3-week PK run-in period as an I.V. infusion at a dose of 75 mg/m2
  Treatment Cycles: Cisplatin administered on Day 1 of every 3-week cycle as an I.V. infusion at a dose of 75 mg/m2

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (PK) of necitumumab in combination with gemcitabine-cisplatin in participants with advanced malignant solid tumors and to assess the potential for drug-drug interactions between necitumumab and gemcitabine-cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Have documented advanced or metastatic malignant solid tumors (except for colorectal tumors with KRAS mutation) that are resistant to standard therapy or for which no standard therapy is available
* May have measurable or non-measurable disease
* Have resolution to Grade 0 or 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE 4.0) of all clinically significant toxic effects (other than alopecia) of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1
* Have adequate hepatic, hematologic and renal function
* If female, are surgically sterile, postmenopausal, or agree to be compliant with a highly effective contraceptive method during and for 6 months after the treatment period. If male, are surgically sterile or agree to be compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period
* Female participants of childbearing potential have a negative serum pregnancy test within 7 days prior to the first dose of study therapy

Exclusion Criteria:

* Have received a systemic anticancer agent (including EGFR tyrosine kinase inhibitors) or device within 28 days prior to first dose of study therapy
* The most recent anticancer therapy received by the participant included either gemcitabine or cisplatin (or both)
* Have received radiotherapy within 14 days prior to first dose of study therapy
* Have received cytotoxic chemotherapy within 21 days prior to first dose of study therapy
* Are receiving concurrent treatment with another anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy, radiation therapy, chemoembolization, or targeted therapy
* Are considered surgical candidates (with resectable disease)
* Have brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants
* Have narrowing of or blockage in large veins
* Have coronary artery disease or uncontrolled congestive heart failure
* Have uncontrolled angina pectoris, or experienced myocardial infarction within 6 months prior to first dose of study therapy
* Have an ongoing or active infection (requiring treatment), including active tuberculosis or known infection with the human immunodeficiency virus
* Have a history of significant neurological or psychiatric disorders, including dementia, seizures, or bipolar disorder
* Have known drug or alcohol abuse
* If female, are pregnant or breastfeeding
* Have had major surgery within 28 days prior to first dose of study medication or subcutaneous venous access device implantation within 7 days prior to first dose of study therapy
* Are currently enrolled in, or discontinued within the 30 days prior to first dose of study therapy from a clinical trial involving an investigational product or nonapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 1 'completers' completed the PK run-in period (3 Weeks) and Cycle 1, Day 1 and Cohort 2 'completers' completed the PK run-in period.
Groups:
- Necitumumab Cohort 1: Necitumumab administered on Day 3 of the 3-week PK run-in period as an intravenous (IV) infusion at an absolute dose of 800 milligrams (mg). Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
  Participants in Cohort 1 received necitumumab Process C drug product. Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/square meter (m2).
  Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
- Necitumumab Cohort 2: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg. Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
  Participants in Cohort 2 received necitumumab drug product manufactured using a new and comparable necitumumab drug substance (Process D drug product).
  Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/m2.
  Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
Period: Overall Study
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Started | 18 | 17
Received at Least 1 Dose of Study Drug | 18 | 17
Completed | 15 | 17
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Progressive Disease | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Necitumumab Cohort 1; Necitumumab Cohort 2: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg. Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
  Participants in Cohort 1 received necitumumab Process C drug product and participants in Cohort 2 received necitumumab Process D drug product.
  Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/m2.
  Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
- Total: Total of all reporting groups
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2 | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (15.54) | 58.2 (13.84) | 56.7 (14.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 17 | 14 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline [Number; unit: participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). 0 - Fully Active. 1 - Ambulatory, Restricted Strenuous Activity. 2 - Ambulatory, No Work Activities. 3 - Partially Confined to Bed, Limited Self Care. 4 - Completely Disabled. 5 - Death.
  participants
    0 | 9 | 7 | 16
    1 | 9 | 10 | 19
    >=2 | 0 | 0 | 0
Disease Characteristics - Tumor Type [Number; unit: participants]
  Breast Carcinoma | 3 | 4 | 7
  Ovarian Carcinoma | 2 | 1 | 3
  Small Cell Lung Carcinoma | 2 | 1 | 3
  Thymic Tumor | 2 | 0 | 2
  Nonsmall Cell Lung Carcinoma | 2 | 0 | 2
  Melanoma | 1 | 1 | 2
  Head and Neck Carcinoma | 1 | 1 | 2
  Endometrial Carcinoma | 1 | 1 | 2
  Hepatobilliary Carcinoma | 1 | 0 | 1
  Left Parotid | 1 | 0 | 1
  Liver | 1 | 0 | 1
  Granulosa Cell Tumor of the Ovary | 1 | 0 | 1
  Mesothelioma | 0 | 1 | 1
  Neuroendocrine Tumor | 0 | 1 | 1
  Hepatocellular Carcinoma | 0 | 1 | 1
  Esophageal Carcinoma | 0 | 1 | 1
  Colorectal Carcinoma | 0 | 1 | 1
  Sarcoma, soft tissue | 0 | 1 | 1
  Adenocarcinoma of the Ampula of Vater | 0 | 1 | 1
  Pancreatic Carcinoma | 0 | 1 | 1
Prior Anti-Cancer Therapy [Number; unit: participants] — Not all participants received prior anti-cancer therapy.
  participants
    Any Prior Radiotherapy | 13 | 10 | 23
    Any Prior (Adjuvant/Neoadjuvant) Systemic Therapy | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Necitumumab
Time Frame: Run-In Period Day 3 Cohort 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 Hour (h) Post Start of Infusion; Cycle 1, Day 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion
Population: All participants who received at least one dose of study drug and had evaluable data for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Groups:
- Necitumumab Cohort 1 Day 3 Run-in: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg. Participants in Cohort 1 received necitumumab Process C drug product.
- Necitumumab Cohort 1 Day 1, Cycle 1, Combination: Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg. Participants in Cohort 1 received necitumumab Process C drug product.
Arm/Group | Necitumumab Cohort 1 Day 3 Run-in | Necitumumab Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 18 | 12
microgram/milliliter (ug/mL) | 277 (22) | 315 (23)

2. Primary Outcome: PK: Dose-Normalized Cmax of Gemcitabine
Time Frame: Run-In Period Day 1 Cohort 1: 0,0.5,1,1.5,3,4,6.67 and 24h Post Start of Infusion; Cycle 1, Day 1: 0, 0.50, 1, 1.5, 3, 4.67, 6.67 and 24 h Post Start of Infusion
Population: All participants who received at least one dose of study drug and had evaluable data for PK. Per protocol, no data were collected for this assessment for participants in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram(ng)/mL/mg
Groups:
- Gemcitabine Cohort 1 Day 1 PK Run-In: Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/m2.
- Gemcitabine Cohort 1 Day 1, Cycle 1, Combination: Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
Arm/Group | Gemcitabine Cohort 1 Day 1 PK Run-In | Gemcitabine Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 18 | 12
nanogram(ng)/mL/mg | 4.83 (66) | 7.87 (43)

3. Primary Outcome: PK: Dose-Normalized Cmax of Cisplatin
Time Frame: Run-In Period Day 1 Cohort 1: 0, 2, 2.03, 2.25, 3, 3.67 and 5.67 h Post Start of Infusion; Cycle 1, Day 1: 0, 2, 2.03, 2.25, 3, 3.67 and 5.67 h Post Start of Infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/mL/mg
Groups:
- Cisplatin Cohort 1 Day 1 Run-in: Cisplatin administered on Day 1 of the 3-week PK run-in period as an IV infusion of 75 mg/m2.
- Cisplatin Cohort 1 Day 1, Cycle 1, Combination: Cisplatin administered 75 mg/m2 on Days 1 and 8 of every 3-week cycle as an IV infusion.
Arm/Group | Cisplatin Cohort 1 Day 1 Run-in | Cisplatin Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 18 | 12
nanogram (ng)/mL/mg | 19.2 (21) | 22.1 (30)

4. Primary Outcome: PK: Area Under Concentration-Time Curve From Zero to Time 168 (AUC[-168]) of Necitumumab
Time Frame: Run-In Period Day 3 Cohort 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion; Cycle 1, Day 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hour(h)/mL
Groups:
- Necitumumab Cohort 1 Day 3 Run-In: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg.
- Necitumumab Cohort 1 Day 1, Cycle 1, Combination: Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
Arm/Group | Necitumumab Cohort 1 Day 3 Run-In | Necitumumab Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 18 | 11
ug*hour(h)/mL | 21900 (24) | 22900 (34)

5. Secondary Outcome: Number of Participants With Anti-Necitumumab Antibodies
Description: A participant was considered to have an anti-necitumumab antibody response if anti-drug antibodies (ADA) were confirmed positive. Treatment emergent antibodies were defined as any anti-necitumumab antibody titer equal to or greater than 4-fold the participant's baseline titer.
Time Frame: Baseline through, 30-Day Follow-Up
Population: All participants who received at least one dose of study drug and had evaluable baseline and postbaseline data for antibodies.
Measure: Number; unit: participants with immunogenicity samples
Groups:
- Necitumumab Cohort 1: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg. Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
  Participants in Cohort 1 received necitumumab Process C drug product. Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/m2.
  Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
- Necitumumab Cohort 2: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg. Necitumumab administered on Days 1 and 8 of every 3-week cycle as an IV infusion at an absolute dose of 800 mg.
  Participants in Cohort 2 received necitumumab Process D drug product.
  Gemcitabine administered on Day 1 of the 3-week PK run-in period as an IV infusion at a dose of 1250 mg/m2.
  Gemcitabine administered on Days 1 and 8 of every 3-week cycle as an IV infusion at a dose of 1250 mg/m2.
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Number analyzed (Participants) | 18 | 17
participants with immunogenicity samples
  ADA Positive | 3 | 0
  TE Antibodies | 1 | 0
  Neutralizing Antibodies | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR]) (Antitumor Activity of Necitumumab in Combination With Gemcitabine-cisplatin Chemotherapy)
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.1, CR was defined as the disappearance of all target and non-target lesions; PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD. Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence)/total number of participants treated) * 100.
Time Frame: Baseline to Measured Progressive Disease (Up to 14 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Number analyzed (Participants) | 18 | 17
percentage of participants | 16.7 [3.6 to 41.4] | 5.9 [0.1 to 28.7]

7. Secondary Outcome: PK: Cmax of Necitumumab After Administration of Process C and Process D Drug Product
Time Frame: Run-In Period Day 3 Cohort 1 and Cohort 2: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion
Population: All participants who received at least one dose of study drug and had evaluable data for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Number analyzed (Participants) | 18 | 17
ug/mL | 277 (22) | 300 (36)

8. Primary Outcome: PK: Dose-Normalized AUC(0-24) of Gemcitabine
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Gemcitabine Cohort 1 Day 1 PK Run-in | Gemcitabine Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 17 | 9
ng*h/mL/mg | 2.71 (45) | 3.31 (33)

9. Secondary Outcome: PK: AUC(0-∞) of Necitumumab After Administration of Process C and Process D Drug Product
Time Frame: Run-In Period Day 3 Cohort 1 and Cohort 2: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion
Population: All participants who received at least one dose of study drug and had evaluable data for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Number analyzed (Participants) | 14 | 14
ug*h/mL | 33800 (33) | 35500 (35)

10. Primary Outcome: PK: Dose-Normalized AUC(0-5) of Cisplatin
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Cisplatin Cohort 1 Day 1 Run-in | Cisplatin Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 17 | 12
ng*h/mL/mg | 61.5 (20) | 67.3 (24)

11. Primary Outcome: PK: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity, (AUC[0-∞]) of Necitumumab
Time Frame: Run-In Period Day 3 Cohort 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion; Cycle 1 Day 1: 0, 0.83, 1.33, 1.83, 3.83, 7.5, 24.83, 72 and 168 h Post Start of Infusion
Population: All participants who received at least one dose of study drug and had evaluable data for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Groups:
- Necitumumab Cohort 1 Day 3 PK Run-In: Necitumumab administered on Day 3 of the 3-week PK run-in period as an IV infusion at an absolute dose of 800 mg.
Arm/Group | Necitumumab Cohort 1 Day 3 PK Run-In | Necitumumab Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 14 | 8
ug*h/mL | 33800 (33) | 26400 (30)

12. Primary Outcome: PK: Dose Normalized AUC(0-∞) of Gemcitabine
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Gemcitabine Cohort 1 Day 1 PK Run-in | Gemcitabine Cohort 1 Day 1, Cycle 1, Combination
Number analyzed (Participants) | 17 | 9
ng*h/mL/mg | 2.72 (45) | 3.32 (33)

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Necitumumab Cohort 1 | Necitumumab Cohort 2
Serious Adverse Events (participants affected / at risk) | 5/18 | 8/17
Other Adverse Events (participants affected / at risk) | 18/18 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab Cohort 1 (N=18) | Necitumumab Cohort 2 (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Necitumumab Cohort 1 (N=18) | Necitumumab Cohort 2 (N=17)
Anaemia (Blood and lymphatic system disorders) | 10 (51) | 13 (50)
Anisocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (8) | 5 (14)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (10)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (25) | 9 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (25) | 6 (26)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Growth of eyelashes (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 3 (3)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (13)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (15) | 10 (26)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (13) | 6 (16)
Asthenia (General disorders) | 1 (2) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 3 (4)
Device deployment issue (General disorders) | 1 (1) | 0 (0)
Device leakage (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 14 (19) | 13 (28)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Implant site erythema (General disorders) | 1 (1) | 0 (0)
Implant site irritation (General disorders) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (5)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (4)
Tenderness (General disorders) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (2) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (4) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (6)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 6 (7)
Alanine aminotransferase decreased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (15) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 11 (16) | 8 (12)
Blood albumin decreased (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (9) | 2 (5)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 4 (11) | 5 (15)
Blood fibrinogen increased (Investigations) | 2 (2) | 2 (2)
Blood magnesium decreased (Investigations) | 3 (3) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 4 (9) | 3 (3)
Blood uric acid increased (Investigations) | 0 (0) | 1 (2)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Carbohydrate antigen 125 increased (Investigations) | 1 (1) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 0 (0) | 2 (2)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 1 (1)
Fibrin d dimer increased (Investigations) | 5 (6) | 2 (3)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 3 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (5) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (13) | 5 (22)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 3 (3) | 0 (0)
Monocyte count increased (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (24) | 4 (12)
Neutrophil count increased (Investigations) | 5 (5) | 0 (0)
Platelet count decreased (Investigations) | 8 (13) | 5 (15)
Platelet count increased (Investigations) | 3 (3) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 2 (2)
Prothrombin time prolonged (Investigations) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 2 (4) | 0 (0)
Urine leukocyte esterase (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 4 (4)
Weight increased (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 10 (23) | 7 (15)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (12) | 9 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6) | 5 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (20) | 7 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (30) | 12 (32)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7) | 4 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2) | 7 (10)
Headache (Nervous system disorders) | 4 (6) | 5 (7)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 3 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (7)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 1/11 (1) | 0/10 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (8)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (10) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days